CLINICAL TRIAL: NCT01246505
Title: Peripheral Facilitated Antegrade Steering Technique in Chronic Total Occlusions
Acronym: PFAST-CTOs
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: BridgePoint Medical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200-0012
Record Dates: First submitted 2010-11-19; First posted 2010-11-23 (Estimated); Last update posted 2012-07-12 (Estimated); Status verified 2012-07

CONDITIONS: Chronic Total Occlusion
MeSH Terms: interventions — Angioplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: CTO Crossing and Percutaneous transluminal angioplasty — Crossing of the CTO with the BridgePoint Medical System and subsequent treatment of the CTO via PTA (specific devices to be used for PTA at investigators' discretion)

SUMMARY:
Study of the BridgePoint Medical System in the crossing of chronic total occlusions of the lower extremities.

ELIGIBILITY:
Inclusion Criteria:

* suitable candidate for non-emergent, peripheral angioplasty
* documented de-novo or restenotic peripheral CTO lesion with TIMI 0 flow for at least 90 days and satisfactory distal vessel visualization (collateral supply)
* limb ischemia or claudication, Rutherford class I-III (grade 1-5) caused by the occluded artery

Exclusion Criteria:

* intolerance to aspirin or a neutropenic response to Ticlopidine or Clopidogrel
* appearance of thrombus or intraluminal filling defects
* peripheral intervention in the target limb within two weeks of the procedure
* renal insufficiency (serum creatinine of > 2.3 mg/dl)
* contraindication to a peripheral artery intervention
* participation in another investigational protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2011-07; Primary Completion 2011-12 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Incidence of Patients with a Major Adverse Events (MAE) | 30 Day
  MAE is defined as death, major unplanned amputation, perforation requiring intervention, or target lesion revascularization due to complication.
Incidence of Intraprocedural Technical Success | Intraprocedural (<24 hours)
  Technical success is defined as the placement of a guidewire in the true lumen distal to the CTO

CONTACTS AND LOCATIONS:
Overall Officials: William A Gray, MD, Principal Investigator — Columbia University
Locations (10):
- United States (10):
  - St. Luke's Medical Center, Phoenix, Arizona
  - University of Southern California Medical Center, Los Angeles, California
  - Torrance Memorial Medical Center, Torrance, California
  - University of Colorado Denver, Denver, Colorado
  - Emory University Medical Center, Atlanta, Georgia
  - Prairie Cardiovascular Consultants, Springfield, Illinois
  - Columbia University Medical Center, New York, New York
  - Wake Heart Center, Raleigh, North Carolina
  - Dallas VA Medical Center, Dallas, Texas
  - St. Joseph Hospital, Bellingham, Washington